CLINICAL TRIAL: NCT02089204
Title: Clinical Feasibility Study of Hypoxia Imaging -Guided IMRT on the Individualized Radiotherapy of Nasopharyngeal Carcinoma
Brief Title: Hypoxia Imaging -Guided Radiotherapy of Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Xuzhou Medical University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Longzhen Zhang, MD,Professor, Xuzhou Medical University
Other Study IDs: H201021
Record Dates: First submitted 2014-03-09; First posted 2014-03-17 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Hypoxia Imaging -Guided Radiotherapy; PET/CT; simultaneous modulated accelerated radiation therapy (SMART)
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- FMISO-PET/CT: 18F-MISO PET/CT -guided dose escalation chemoradiotherapy. All patients were given concurrent chemoradiotherapy within two weeks of diagnosis. Radiotherapy was delivered using the simultaneous modulated accelerated radiation therapy (SMART) IMRT technique in the dose-escalation treatment arms. Concurrent chemotherapy consisted of cisplatin (20mg / m2 ,iv, d1- 4) and docetaxel (75mg / m2, d1, d8) administered on the 1st and 4th week of treatment. All patients received adjuvant chemotherapy that ranged from 2 to 4 cycles.
  Interventions: Radiation: FMISO-PET/CT; Radiation: contrast-enhanced CT
- FDG-PET/CT: 18F-FDG PET/CT -guided dose escalation chemoradiotherapy. All patients were given concurrent chemoradiotherapy within two weeks of diagnosis. Radiotherapy was delivered using the simultaneous modulated accelerated radiation therapy (SMART) IMRT technique in the dose-escalation treatment arms. Concurrent chemotherapy consisted of cisplatin (20mg / m2 ,iv, d1- 4) and docetaxel (75mg / m2, d1, d8) administered on the 1st and 4th week of treatment. All patients received adjuvant chemotherapy that ranged from 2 to 4 cycles.
  Interventions: Radiation: FDG-PET/CT; Radiation: contrast-enhanced CT
- contrast-enhanced CT: contrast-enhanced CT -guided dose escalation chemoradiotherapy . GTVs were delineated based on fusing diagnostic CT images with simulation CT images.All patients were given concurrent chemoradiotherapy within two weeks of diagnosis. Radiotherapy was delivered using the simultaneous modulated accelerated radiation therapy (SMART) IMRT technique in the dose-escalation treatment arms. Concurrent chemotherapy consisted of cisplatin (20mg / m2 ,iv, d1- 4) and docetaxel (75mg / m2, d1, d8) administered on the 1st and 4th week of treatment. All patients received adjuvant chemotherapy that ranged from 2 to 4 cycles.
  Interventions: Radiation: contrast-enhanced CT

INTERVENTIONS:
Radiation: FMISO-PET/CT — Fluorine-18-labeled fluoromisonidazole PET/CT-guided dose escalation chemoradiotherapy (group C). Radiotherapy was delivered using the simultaneous modulated accelerated radiation therapy (SMART) technique in the dose-escalation treatment arms. Patients received concurrent and adjuvant chemotherapy.
  Other Names: fluorine-18-labeled fluoromisonidazole
  Groups: FMISO-PET/CT
Radiation: FDG-PET/CT — 18F-FDG PET/CT -guided dose escalation chemoradiotherapy. Radiotherapy was delivered using the simultaneous modulated accelerated radiation therapy (SMART) technique in the dose-escalation treatment arms. Patients received concurrent and adjuvant chemotherapy.
  Other Names: fluorine-18 deoxyglucose
  Groups: FDG-PET/CT
Radiation: contrast-enhanced CT — contrast-enhanced CT -guided dose escalation chemoradiotherapy. Radiotherapy was delivered using the simultaneous modulated accelerated radiation therapy (SMART) technique in the dose-escalation treatment arms. Patients received concurrent and adjuvant chemotherapy

SUMMARY:
Nasopharyngeal carcinoma (NPC) differs from other head and neck malignancies in terms of its epidemiology, pathology, and treatment outcome . It is endemic in China and is one of the major public health problems. Concurrent radiotherapy and chemotherapy is the primary treatment for patients with NPC. Despite such aggressive treatment, many patients with locally advanced NPC still develop locally recurrent disease. Since local control is directly related to patient morbidity and mortality in NPC, there is a strong need to identify methods to further improve treatment outcome for NPC.

One strategy to improve local control is to escalate the dose of radiotherapy. This is because local control has been shown to be directly related to the radiotherapy dose. Several different techniques, including brachytherapy, stereotactic radiosurgery, and dose-painting intensity modulated radiotherapy (IMRT), have been used to increase radiotherapy dose. However, due to the large number of critical anatomic structures near the nasopharynx, dose-escalation in NPC can also lead to increased toxicities. One technique that has achieved dose-escalation with minimal increase in toxicity is simultaneous modulated accelerated radiation therapy (SMART). The main challenge for such treatment is to identify the appropriate tumor volume to receive the high-dose radiotherapy. Conventional dose-escalation is conducted using computed tomography (CT) to identify the gross tumor volume (GTV). However, recent progress with F-18 fluorodeoxyglucose positron emission tomography/computed tomography (18F-FDG-PET/CT) in treatment planning allows more accurate tumor volume delineation. We hypothesize that the use of PET/CT in treatment planning can improve dose-escalation radiotherapy for NPC which in turn can improve therapeutic efficacy while reducing toxicity. PET/CT imaging of tissue hypoxia using [F-18]fluoromisonidazole (FMISO), the most widely used nitroimidazole imaging agent.Given that there has been no clinical trials directly comparing conventional chemoradiotherapy to CT-guided dose-escalation chemoradiotherapy or PET/CT guided dose-escalation chemoradiotherapy in locally advanced NPC.This was a study to evaluate the role of FMISO-PET hypoxia imaging for predicting survival in NPC,our study aims to compare the local control, overall survival and toxicities of the three treatment regimens..

DETAILED DESCRIPTION:
Study Design Patients with previously untreated Stages III~IVA (AJCC 6th Edition) of locally advanced NPC, Karnofsky performance status≥70, and good bone marrow, liver and kidney functions (white blood count ≥ 4.0×109/L, platelets ≥ 100×109/L, albumin ≥30 g/L , creatinine ≤100μmol/L) were enrolled on this study. Patients younger than 18, those with a prior (within 5 years) or synchronous malignancy were excluded. Pretreatment evaluations consisted of a history and physical, dental and laboratory studies. The clinical stage was determined based on all information provided by examinations including contrast enhanced CT and magnetic resonance imaging (MRI) of head and neck, Chest X-ray, liver sonography, bone scan, and 18F-FDG-PET. All tumors were histologically confirmed except those of distant sites.

Patients who met the eligibility criteria were randomized 1:1:1 into the three treatment arms: conventional chemoradiotherapy (group A), FDG PET/CT -guided dose escalation chemoradiotherapy (group B) and FMISO PET/CT -guided dose escalation chemoradiotherapy (group C). All patients were given concurrent chemoradiotherapy within two weeks of diagnosis. Radiotherapy was delivered using the simultaneous modulated accelerated radiation therapy (SMART) IMRT technique in the dose-escalation treatment arms. Concurrent chemotherapy consisted of cisplatin (20mg / m2 ,iv, d1- 4) and docetaxel (75mg / m2, d1, d8) administered on the 1st and 4th week of treatment. All patients received adjuvant chemotherapy that ranged from 2 to 4 cycles.

Follow-up and statistical analysis Planned patient assessment included physical examination and fiberoptic nasopharyngoscopy every 3 months to 3 years starting at 4 weeks post-treatment. A contrast-enhanced CT or MRI of the head and neck is also obtained at each follow up. After 3 years, the patients were followed yearly thereafter. Suspected recurrences were histologically proven. To assess for distant metastasis, CT of the chest and bone scan were obtained every half a year. During every follow-up visit, treatment toxicity were assessed. Radiotherapy-related toxicities were graded according to the Acute and the Late Radiation Morbidity Scoring Criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Chemotherapy-related toxicities (except nausea or alopecia) were graded by the criteria of the WHO.

All events were measured from the date of randomization. OS was defined as the time from the date of radiotherapy to death or the latest date known to be alive. Durations were calculated from the end of treatment. The Kaplan-Meier method was used to calculate the actuarial rates of local control, DFS and OS. The χ2 test was used for comparing incidence rates and categorical variables and Student's t-test was used for comparing the means of continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed NPC by biopsy,
* no evidence of distant metastasis,
* no previous treatment for NPC,
* Stages III~IVA (AJCC 7th Edition) of locally advanced ,
* adequate liver function (albumin ≥30 g/L),
* adequate renal function (creatinine ≤100μmol/L) ,
* adequate bone marrow function(white blood count ≥ 4.0×109/L, platelets ≥ 100×109/L),
* Karnofsky performance status≥70,

Exclusion Criteria:

* Patients younger than 18,
* those with a prior (within 5 years) or synchronous malignancy were excluded.
* presence of distant metastases,
* pregnancy or lactation,
* other concomitant malignant disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between June 2010 to June 2015, patients from Department of Radiation Oncology, Affiliated Hospital of Xuzhou Medical College.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
local progression-free (LPF) survival rates | 5 years
  LPF was defined as the time from the date of radiotherapy to local progression in the five years after treatment.Durations were calculated from the end of treatment.

SECONDARY OUTCOMES:
disease-free survival (DFS) | 5 years
  DFS was defined as the time from the date of radiotherapy to recurrence or local progression in the five years after treatment.Durations were calculated from the end of treatment.
overall survival (OS) | 5 years
  OS was defined as the time from the date of radiotherapy to death or the latest date known to be alive. Durations were calculated from the end of treatment.

OTHER OUTCOMES:
acute toxicities | from treatment start to 4 weeks post-treatment
  Acute toxicities were mucositis, nausea/vomiting, arrest of bone marrow, skin desquamation.
  Radiotherapy-related toxicities were graded according to the Acute and the Late Radiation Morbidity Scoring Criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Chemotherapy-related toxicities (except nausea or alopecia) were graded by the criteria of the WHO.
Late toxicities | from 4 weeks post-treatment to 5 years.
  Late toxicities were skin dystrophy, subcutaneous fibrosis, xerostomia, and hearing loss.
  Radiotherapy-related toxicities were graded according to the Acute and the Late Radiation Morbidity Scoring Criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Chemotherapy-related toxicities (except nausea or alopecia) were graded by the criteria of the WHO.

CONTACTS AND LOCATIONS:
Overall Officials: ZHANG Longzhen, MD, Study Chair — Xuzhou Medical University; Wang Andrew Z., MD and PHD, Study Director — University of North Carolina at Chapel Hill, USA; Wang Jianshe, M.M., Principal Investigator — Xuzhou Medical University; Xin Yong, M.M., Principal Investigator — Xuzhou Medical University; Xu Kai, MD, Principal Investigator — Xuzhou Medical University; Tang Tianyou, M.M., Principal Investigator — Xuzhou Medical University; Ding Xin, M.M., Principal Investigator — Xuzhou Medical University

REFERENCES:
- [Derived] Wang J, Zheng J, Tang T, Zhu F, Yao Y, Xu J, Wang AZ, Zhang L. A Randomized Pilot Trial Comparing Position Emission Tomography (PET)-Guided Dose Escalation Radiotherapy to Conventional Radiotherapy in Chemoradiotherapy Treatment of Locally Advanced Nasopharyngeal Carcinoma. PLoS One. 2015 Apr 27;10(4):e0124018. doi: 10.1371/journal.pone.0124018. eCollection 2015. PMID 25915944